CLINICAL TRIAL: NCT01267630
Title: The Validity and Reliability of Thai Version of the Confusion Assessment Method for the Intensive Care Unit (CAM -ICU)
Brief Title: The Validity of the Thai Version of the Confusion Assessment Method
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chiang Mai University (Other)
Responsible Party: Tanyong Pipanmekaporn, Department of Anesthesiolgy, Faculty of Medicine, Chiang Mai University. Chiang Mai, Thailand, 50200
Other Study IDs: ANE100806A11; ANE10-08-06A-11 (Other: Ethic committee, Faculty of Medicine, Chiang Mai University)
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-01

CONDITIONS: Delirium
Keywords: Delirium of Mixed Origin; Subacute Delirium; Mental Disorders, Organic; Organic Brain Syndrome, Nonpsychotic; Organic Mental Disorders; Organic Mental Disorders, Psychotic; Psychoses, Traumatic; Cognition Disorder; Confusion state; Disorientation
MeSH Terms: conditions — Delirium; Neurocognitive Disorders; Cognition Disorders; Confusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical ICU: Patients are admitted to the surgical ICU of Chiang Mai University Hospital within 48 hours .

SUMMARY:
The purpose of this study is to determine the validity and reliability of the Thai version of the Confusion Assessment Method for the intensive care (CAM-ICU) in the elderly and the prevalence of delirium in elderly.

DETAILED DESCRIPTION:
The incidence of delirium in intensive care unit varied between 20 and 80% depending on many factors such as types of study, diagnostic tools, severity of patients.The occurrence of delirium is common in elderly patients. However, the prevalence of delirium in the intensive care has not been reported in Thailand. There is no common tool used for detecting delirium in Thai ICU. Currently, CAM-ICU has been developed for nonpsychiatric physician and other health care professionals to detect delirium. The sensitivity and specificity of CAM-ICU was 91-93% and 89-100% respectively. In addition, it has been translated to many version to diagnose deliriums for all over the world. In Thailand, there is no common tool used for detecting delirium in ICU. The use of CAM-ICU may be useful in Thai ICU settings.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 55 years old

Exclusion Criteria:

* Severe visual or auditory impairment
* Comatose or moribund patients
* Unable to communicate with Thai language

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are admitted to the surgical ICU of Chiang Mai University Hospital within 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Thai version of the CAM-ICU for diagnosis of ICU delirium | within 48 hours after admission

SECONDARY OUTCOMES:
The prevalence of elderly delirium patients in intensive care unit | within 48 hours after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Tanyong Pipanmekaporn, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Chiang Mai University , Chiang Mai, Thailand,50200
Locations (3):
- Thailand (3):
  - Chiang Mai University Hospital, Maung, Chiang Mai
  - Department of Anesthesiology, Faculty of Medicine, Maung, Chiang Mai
  - Chiang Mai University Hospital, Muang, Chiang Mai